CLINICAL TRIAL: NCT01472289
Title: To Study and Demonstrate the Safety and Efficacy of RES-Q Prepared Bone Marrow Mononuclear Cells Injected Into Ischemic Tissue of Patients With Non-Reconstructable Critical Limb Ischemia (CLI).
Brief Title: Safety and Efficacy of Autologous Bone Marrow Mononuclear Cells in Patients With Severe Critical Limb Ischemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: TotipotentSC Scientific Product Pvt. Ltd. (Industry)
Collaborators: Thermogenesis Corp. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TPSC/POC/BMSC/CLI/2010/1b; 050343290-0702201132855389 (Registry Identifier: Clinical Trials Registry - India (CTRI))
Record Dates: First submitted 2011-07-18; First posted 2011-11-16 (Estimated); Results first posted 2015-11-18 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-10

CONDITIONS: Critical Limb Ischemia
Keywords: CLI; Peripheral arterial disease
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BMMNC treated group (Experimental): Autologous bone marrow mononuclear cell concentrate (BMMNCs) prepared using the Res-Q 60 technology (a point of care system) to be injected intramuscularly into multiple sites in the ischemic muscle tissue of the affected limb at 0.5 cc/injection for a total of 15-20 cc.
  Interventions: Other: Autologous Bone Marrow Mononuclear cells (BMMNCs)

INTERVENTIONS:
Other: Autologous Bone Marrow Mononuclear cells (BMMNCs) — Multiple intramuscular injections of concentrated bone marrow derived mononuclear cells (0.5 cc/injection) into the ischemic muscle of the affected limb.
  Other Names: Autologous bone marrow mononuclear cell concentrate

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the concentrated autologous bone marrow derived stem cells for the treatment of Critical Limb Ischemia patients.

DETAILED DESCRIPTION:
A total of 15 patients suffering from end stage IV and V Rutherford /CLI in whom all previous therapeutic strategies failed (e.g. surgical revascularization) will be selected and undergo local transplantation of autologous BMMNCs. Conventional treatments include angioplasty and /or bypass to remove blood vessel blockage for restoring blood supply, along with prescribed medicines that aid in ulcer recovery and wound healing and debridement of damaged/infected tissue. Amputation is inevitable in many cases because some blood capillaries cannot be corrected and restenosis of vessels is very common. Cell therapies with mononuclear cells from patients own bone marrow is promising because these stem cells are capable of stimulating and regenerating capillaries and blood vessels (neovascularization).

This is a Phase Ib (feasibility study), prospective, non randomized and open labeled study aimed to find out the safety and efficacy of intramuscular autologous bone marrow mononuclear cells implantation in patients with chronic critical limb ischemia.

The efficacy/safety of this therapy will be assessed by using several endpoints such as (a) prevention of amputation, (b) wound healing and (c) degree of angiogenesis. In order to assess the limb ischemia, the measurements will be performed at pre- and post transplantation at a variety of time intervals. The measurements include: ABI-ankle brachial index, Transcutaneous partial pressure of Oxygen (TcPO2), 6 min walk test, Rest pain and intermittent Claudication assessment, Healing of ulcers/ wounds and angiography of the affected limb.

ELIGIBILITY:
Inclusion Criteria:

* Atherosclerotic ischemic peripheral vascular disease (PVD) or Thromboangiitis Obliterans with severe Critical Limb Ischemia (Rutherford Category 4 and 5: ischemic pain at rest and minor tissue loss and Fontaine Class 4: Ischemic ulcers or gangrene, whivh may be dry or humid).
* A non-surgical candidate for revascularization e.g. prior vascular reconstruction, inability to locate a suitable vein for grafting, diffuse multi- segment disease, or extensive infra-popliteal disease not amenable to a vascular graft.
* Major amputation recommended patients due to severe life threatening PAD.
* Subjects must be on maximal tolerated medical therapy for peripheral vascular disease including A) Cessation of smoking B) Referral to endocrinologist for control of HgA1c to < 8% mg/dl, C) control of hyperlipidemia with statins or other anti-hyperlipidemic drugs as indicated, D) control of hypertension as indicated E) Antiplatelet therapy with aspirin and / or cilostazol (unless medically contraindicated, e.g. bleeding or allergy).
* Ankle Brachial Pressure Index (ABI) ≤ 0.6 or ankle systolic pressure ≤ 60 mm Hg or TcPO2 ≤ 35 mmHg in the foot.
* Subjects who are able to understand the requirements of the study, and willing to provide voluntary written informed consent, which abide by the study requirements, and agree to return for required follow-up visits.

Exclusion Criteria:

* Subjects with CLI suitable for surgical or percutaneous revascularization and Subjects with acute and chronic inflammatory condition.
* CLI patient requiring amputation proximal to trans-metatarsal level
* Subjects with spreading (wet) gangrene
* Subjects with gait disturbance for reasons other than CLI.
* Subjects with poorly controlled diabetes mellitus.
* Subjects diagnosed with Thromboangiitis Obliterans (Buerger's Disease) who are smokers and are unwilling or unable to quit smoking or the physician feels the smoking cessation is doubtful.
* Subjects having moderate to severe COPD with GOLD Classification IIb or III.
* Uncontrolled congestive heart failure or Subjects with left ventricular ejection fraction < 25% or AHA Stage C or D heart failure or NYHA Class IV CHF
* Stroke or myocardial infarction within last 3 months.
* Subjects who are contraindicated for CT Angiogram.
* Illnesses or conditions that are uncontrolled or whose control, in the opinion of the Principal Investigator, may be jeopardized by participation in this study or by the complications of this therapy.
* Documented terminal illness or cancer or any concomitant disease process with a life expectancy of less than 1 year.
* Subjects already enrolled in another investigational drug trial or completed within 3 months.
* History of severe alcohol or drug abuse within 3 months of screening.
* Hb% < 10 gm%; Serum creatinine ≥ 2.0mg%; Serum total bilirubin ≥2.0mg%; HbA1c > 8.0%.
* Women of child bearing potential; pregnant and lactating women.
* Subjects with a) myocardial infarction within the last 30 days or left ventricular ejection fraction < 35%, B) Subjects with a cerebrovascular accident within the last 6 months.
* INR > 1.5 at the time of Bone Marrow harvest.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2011-02; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Venkatesh Ponemone, PhD, Study Director — TotipotentRX, Center for Cellular Medicine; Kenneth Harris, MS, Study Chair — TotipotentRX, Centre for Cellular Medicine; Suhail Bukhari, MBBS, FNBE, Principal Investigator — Fortis Escorts Heart Institute and Research Centre
Locations (1):
- Fortis Escorts Heart Institute & Research Centre, New Delhi, New Delhi, India

RESULTS

PARTICIPANT FLOW:
Groups:
- BMMNC Treated Group: All the subjects enrolled in the study were treated using autologous Bone Marrow Mononuclear Cells (BMMNCs) concentrate prepared using the Res-Q 60 technology (a point of care system) and injected the concentrate intra-muscularly into multiple sites in the ischemic tissue of the affected limb at 0.5 cc/injection for a total of 15-20 cc.
Period: Overall Study
Arm/Group | BMMNC Treated Group
Started | 17
Completed | 15
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: A total of 17 subjects who met the eligibility criteria were enrolled in this study.
Groups:
- BMMNC Treated Group: All the subjects enrolled in the study were treated using autologous Bone Marrow Mononuclear Cells concentrate (BMMNCs) prepared using the Res-Q 60 technology (a point of care system) and injected intra-muscularly into multiple sites in the ischemic muscle of the affected limb at 0.5 cc/injection for a total of 15-20 cc.
Arm/Group | BMMNC Treated Group
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (13.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 17
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  India | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Major Limb Amputation Free Survival Post BMMNC Administration
Description: The Primary objective of this study was to determine the safety of intramuscular administration of concentrated autologous BMMNCs harvested, and processed using the Res-Q 60 technology (a point-of-care system). Safety measurements included close vigilance for major limb amputation free survival at 1, 3, 6 and 12 months post BMMNCs administration and stringent reporting of AEs and SAEs.
Time Frame: 1, 3, 6 and 12 Months
Population: All the safety end points in the study were analyzed on the ITT population. Out of 17 subjects, adverse events were reported for seven subjects. Of the seven subjects, three underwent major amputation, two reported minor amputation, and two died due to cardiac arrest (unrelated death). Furthermore, major limb amputation free survival rate was 14.
Measure: Number; unit: participants
Groups:
- BMMNC Treated Group: All the subjects enrolled in the study were treated using autologous Bone Marrow Mononuclear Cells concentrate (BMMNCs) prepared using the Res-Q 60 technology (a point of care system) and injected intra-muscularly into multiple sites in the ischemic tissue of the affected limb at 0.5 cc/injection for a total of 15-20 cc.
Arm/Group | BMMNC Treated Group
Number analyzed (Participants) | 17
participants
  Major Limb Amputation Free Survival Rate | 14
  Major Amputation | 3
  Minor Amputation | 2
  Unrelated Death | 2
  Total Adverse Events | 7

2. Secondary Outcome: Degree of Angiogenesis Measured by the Number of Collateral Blood Vessels Formed at 12 Months
Description: Measurement of blood supply facilitated by the formation of collateral blood vessels assessed by CT angiography after the procedure.
Time Frame: Baseline and 12 month
Population: Efficacy measures were established by assessing CLI symptoms known to be reliable and valid. The efficacy endpoints were analyzed on per protocol (PP) basis (N=14).
Measure: Mean (Standard Deviation); unit: Number of Vessels
Arm/Group | BMMNC Treated Group
Number analyzed (Participants) | 14
Number of Vessels
  Number of Collateral vessels at Baseline | 2.42 (0.775)
  Number of Collateral vessels at 12 months | 5.59 (1.146)

3. Secondary Outcome: Measurement of Mean Change in Ankle Brachial Index From Baseline to 12 Months
Description: ABI was used to provide a measure of blood flow in the lower limbs. It is the ratio of the blood pressure in the lower limbs to the blood pressure in the upper limbs. Compared to the upper limb, lower blood pressure in the lower limb is an indication of blocked arteries (peripheral vascular disease). The ABI was calculated by dividing the systolic blood pressure at the ankle by the systolic blood pressures in the arm. ABI test was performed at baseline, 1 month, 3 months, 6 months, and 12 months.
Time Frame: Baseline, 1, 3, 6 and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | BMMNC Treated Group
Number analyzed (Participants) | 14
Ratio
  ABI at Baseline | 0.507 (0.0971)
  ABI at 1 Month | 0.612 (0.1653)
  ABI at 3 Months | 0.819 (0.2829)
  ABI at 6 Months | 0.879 (0.2467)
  ABI at 12 Months | 0.696 (0.2650)

4. Secondary Outcome: Measurement of Change in Transcutaneous Oxygen Pressure (TcPO2) From Baseline to 12 Months
Description: TcPO2 was used to assess the partial pressure (tension) of oxygen in the capillaries of tissues of lower limbs. It was measured by applying a special set of electrodes to the skin. These electrodes contain photoelectric sensors capable of detecting the specific wavelengths of radiation emitted by oxygenated versus reduced hemoglobin.
Time Frame: Baseline, 1, 3, 6 and 12 months
Population: The efficacy endpoints were analyzed on per protocol (PP) basis (N=14).
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | BMMNC Treated Group
Number analyzed (Participants) | 14
mmHg
  TcPO2 at Baseline | 14.66 (6.925)
  TcPO2 at 1 Month | 25.10 (11.906)
  TcPO2 at 3 Months | 36.85 (17.892)
  TcPO2 at 6 Months | 34.58 (15.500)
  TcPO2 at 12 Months | 35.75 (17.035)

5. Secondary Outcome: Change in Rest Pain and Intermittent Claudication Assessment From Baseline to 12 Months
Description: Rest pain is a burning sensation felt at rest, usually in the skin of the foot. It is a symptom of critical ischemia due to severe, chronic, and occlusive peripheral arterial disease (PAD). While, Intermittent Claudication is a crampy leg pain that occurs during exercise, especially walking. The pain is due to the insufficient blood flow in the legs (caused by blocked arteries). Intermittent claudication is the most prominent symptom of PAD.
  Both Rest Pain assessment and Intermittent Claudication assessment was performed through Visual Analog Scale or Visual Analogue Scale (VAS). VAS is a psychometric (self-report) response scale that ranges from 0 to 10, where a mark of zero indicates no pain and a mark of 10 indicates worst possible pain.
Time Frame: Baseline, 1, 3, 6 and 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | BMMNC Treated Group
Number analyzed (Participants) | 14
scores on a scale
  Rest Pain Score at Baseline | 2.80 (0.80)
  Rest Pain Score at 1 Month | 1.2 (1.17)
  Rest Pain Score at 3 Months | 0.6 (0.87)
  Rest Pain Score at 6 Months | 0.4 (0.90)
  Rest Pain Score at 12 Months | 0.0 (0.00)
  Intermittent Claudication Pain Score at Baseline | 7.80 (0.97)
  Intermittent Claudication Pain Score at 1 Month | 4.9 (2.22)
  Intermittent Claudication Pain Score at 3 Months | 2.8 (2.61)
  Intermittent Claudication Pain Score at 6 Months | 1.1 (1.44)
  Intermittent Claudication Pain Score at 12 Months | 0.2 (0.58)

6. Secondary Outcome: Clinical Evaluation for the Presence of Ulcer and/or Gangrene in the Affected Limb From Baseline to 12 Months
Description: Evaluation of the integument for ulceration, gangrene and other skin changes in the affected limb was performed at baseline and follow-up visits at 1 month, 3 months, 6 months, and 12 months.The ulceration and gangrene in the affected limb of the subjects was evaluated by visual clinical inspection.
Time Frame: Baseline, 1, 3, 6 and 12 months
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | BMMNC Treated Group
Number analyzed (Participants) | 14
Participants
  Ulcer and/ or Gangrene present at Baseline | 11
  Ulcer and/or Gangrene present at 1 Month | 10
  Ulcer and/or Gangrene present at 3 Months | 6
  Ulcer and/or Gangrene present at 6 Months | 2
  Ulcer and/ or Gangrene present at 12 Months | 0

7. Secondary Outcome: Number of Participants Able to Walk From Baseline to 12 Months as Measured by 6-Minute Walk Test
Description: Subjects were analyzed to see if they were able to walk any distance and the distance covered by patients in 6 minutes was measured to assess the functional changes from baseline. The American Thoracic Society has issued guidelines for the 6-minute walk test (6 MWT). The 6 MWT is safe, easy to administer, well tolerated, and reflects activities of daily living.
Time Frame: Baseline, 1, 3, 6 and 12 months
Population: as for outcome 2
Measure: Number; unit: Participants
Arm/Group | BMMNC Treated Group
Number analyzed (Participants) | 14
Participants
  Subjects able to walk at baseline | 2
  Subjects able to walk at 1 Month | 8
  Subjects able to walk at 3 Months | 9
  Subjects able to walk at 6 Months | 9
  Subjects able to walk at 12 Months | 9

ADVERSE EVENTS:
Time Frame: Adverse events were reported for the duration of the study, that is, from baseline to 12 Months
Arm/Group | BMMNC Treated Group
Serious Adverse Events (participants affected / at risk) | 7/17
Other Adverse Events (participants affected / at risk) | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMMNC Treated Group (N=17)
Major Limb Amputation (Vascular disorders) | 3 (3)
Minor Limb Amputation (Vascular disorders) | 2 (2)
Death (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less